CLINICAL TRIAL: NCT05727657
Title: A Phase 1 Clinical Trial of Satralizumab as a Treatment for Aneurysmal Subarachnoid Hemorrhage
Brief Title: Satralizumab in Aneurysmal Subarachnoid Hemorrhage
Acronym: SASH
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lost support from the drug manufacturer
Sponsor: University of Florida (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCR43615
Record Dates: First submitted 2023-02-03; First posted 2023-02-14 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Delayed Cerebral Ischemia
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — satralizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Satralizumab (Experimental): Subjects will receive satralizumab 120mg subcutaneous Day 0 and Day 14 after enrollment.
  Interventions: Drug: Satralizumab

INTERVENTIONS:
Drug: Satralizumab — 120mg subcutaneous Day 0 and Day 14

SUMMARY:
In this study, satralizumab will be administered to see whether satralizumab is safe in patients with a burst brain aneurysm and if it may prevent strokes in patients with a burst brain aneurysm.

DETAILED DESCRIPTION:
SASH is a prospective single-arm, single-center, open-label Phase 1 trial of satralizumab 120mg subcutaneous Day 0 and Day 14 in subjects with Hunt Hess grade 1-3, Fisher score 3 aneurysmal subarachnoid hemorrhage and an external ventricular drain or lumbar drain. The trial is designed to demonstrate safety and to detect a signal that satralizumab prevents delayed cerebral ischemia in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged ≥18 years) with Hunt Hess Grade 1-3, Fisher score 3 or 3 and 4, aneurysmal subarachnoid hemorrhage within 72 hours of symptom onset (ruptured aneurysm confirmed by CTA, MRA or DSA)
* Must have surgical or endovascular adequate occlusion of the ruptured aneurysm
* Must have external ventricular drain or lumbar drain.
* Female subjects of child-bearing potential must have negative pregnancy test
* Signed informed consent from subject or legally authorized representative
* Able and willing to comply with followup visits
* Women and males of childbearing potential must agree to appropriate methods of contraception during study participation

Exclusion Criteria:

* Evidence for vasospasm or DCI prior to study enrollment
* Hemodynamically unstable pre-enrollment
* Severe or unstable concomitant condition or disease (e.g., known significant neurological deficit, cancer, hematologic or coronary disease), or chronic condition (e.g., liver disease, kidney disease, or psychiatric disorder), that may increase the risk associated with study participation, or may interfere with the interpretation of study results
* Subjects who have received an investigational product or participated in another interventional clinical study within 30 days prior to enrollment.
* Known hypersensitivity to satralizumab and/or other biologics agents
* Serious infection defined as pneumonia, sepsis/septic shock, and neutropenic fever prior to enrollment
* Any previous treatment with IL-6 inhibitory therapy (e.g. tocilizumab), alemtuzumab, total body irradiation or bone marrow transplantation within 6 months prior to baseline.
* Any previous treatment with anti-CD20, anti-CD19, eculizumab, belimumab, interferon, natalizumab, glatiramer acetate, fingolimod, teriflunomide or dimethyl fumarate within 6 months prior to baseline.
* Any previous treatment with anti-CD4, cladribine or mitoxantrone within 2 years prior to baseline
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 3 months after the final dose of satralizumab
* Women of childbearing potential must have a negative serum pregnancy test result prior to initiation of study drug.
* Any surgical procedure (except for minor surgeries) within 4 weeks prior to baseline.
* Evidence of other demyelinating disease or progressive multifocal leukoencephalopathy (PML).
* Evidence of serious uncontrolled concomitant diseases that may preclude patient participation, such as: other nervous system disease, cardiovascular disease, hematologic/hematopoiesis disease, respiratory disease, muscular disease, endocrine disease, renal/urologic disease, digestive system disease, congenital or acquired severe immunodeficiency.
* Known active infection (excluding fungal infections of nail beds or caries dentium) within 4 weeks prior to baseline.
* History of diverticulitis that, in the Investigator's opinion, may lead to increased risk of complications such as lower gastrointestinal perforation.
* Evidence of active or untreated latent tuberculosis (TB; excluding patients receiving chemoprophylaxis for latent TB infection).
* Evidence of active interstitial lung disease
* Receipt of any live or live attenuated vaccine within 6 weeks prior to baseline and throughout the duration of the study.
* History of malignancy within the last 5 years, including solid tumors, hematologic malignancies and in situ carcinoma (except basal cell and squamous cell carcinomas of the skin, or in situ carcinoma of the cervix uteri that have been completely excised and cured).
* Laboratory exclusion criteria (at screening):
* White blood cells (WBC) <3.0 x103/μL
* Absolute neutrophil count (ANC) <2.0 x103/μL
* Absolute lymphocyte count <0.5 x103/μL
* Platelet count <10 x 104/μL
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 times the upper limit of normal (ULN).
* Patient with known medical history at screening listed for the following must be excluded from this trial:
* Evidence of chronic active hepatitis B (HBV)
* Evidence of chronic active hepatitis C (HCV)
* Positive for hepatitis C virus (HCV) antigen
* Positive for hepatitis B surface antigen (HBsAg)
* Known HIV infection.
* Viral antigen tests for HBV, HCV and HIV to be performed on Day 0 (day of first dose of satralizumab). If the result of HBV, HCV, or HIV comes back positive the 2nd dose of satralizumab (Day 14) will not be administered
* Illicit drug or alcohol abuse within 12 months prior to screening, in the investigator's judgment
* Poor peripheral venous access
* Serious infection requiring oral or IV antibiotics prior to screening
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
* History or presence of an abnormal ECG that is clinically significant in the investigator's opinion, including complete left bundle branch block, second- or third degree atrioventricular heart block, or evidence of prior myocardial infarction

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with elevation of liver transaminases | baseline up to 21 days
  Elevation of liver transaminase (ALT, AST) is defined as >5x upper limit of normal.
Number of participants with neutropenia | baseline up to 21 days
  Neutropenia is defined as neutrophil count below 1 x 10^9/L.
Number of participants with decreased platelet count | baseline up to 21 days
  Decreased platelet count is defined as a platelet count below the lower institutional limit of normal.
Frequency of observed and reported adverse events | baseline up to 90 days following the last administration of study treatment or study discontinuation/termination, whichever is earlier
  An adverse event will be defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational medicinal product (IMP) or other protocol-imposed intervention, regardless of attribution.
Frequency of death | baseline up to 90 days following the last administration of study treatment or study discontinuation/termination, whichever is earlier
  All deaths that occur during the protocol-specified AE reporting period, regardless of attribution, will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Hoh, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida (UF) Health Shands Hospital, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No